CLINICAL TRIAL: NCT01767610
Title: Open-label, Randomized, Repeated Dosing Crossover Study to Evaluate the Pharmacokinetic Interaction Between Micronized Fenofibrate and Pitavastatin in Healthy Adult Subjects
Brief Title: Evaluation of Pharmacokinetic Interaction Between Micronized Fenofibrate and Pitavastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HL-PIF-101
Record Dates: First submitted 2013-01-11; First posted 2013-01-14 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Healthy Male Volunteers
MeSH Terms: interventions — Fenofibrate; pitavastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- micronized fenofibrate (Experimental)
  Interventions: Drug: micronized fenofibrate 160mg
- pitavastatin Ca (Experimental)
  Interventions: Drug: pitavastatin Ca 2mg
- micronized fenofibrate plus pitavastatin Ca (Experimental)
  Interventions: Drug: micronized fenofibrate 160mg plus pitavastatin Ca 2mg

INTERVENTIONS:
Drug: micronized fenofibrate 160mg
  Other Names: Lipilfen cap. 160mg : once daily for 5 days
  Arms: micronized fenofibrate
Drug: pitavastatin Ca 2mg
  Other Names: Livalo tab. 2mg : once daily for 5 days
  Arms: pitavastatin Ca
Drug: micronized fenofibrate 160mg plus pitavastatin Ca 2mg
  Other Names: Lipilfen cap. 160mg plus Livalo tab. 2mg : once daily for 5 days
  Arms: micronized fenofibrate plus pitavastatin Ca

SUMMARY:
To evaluate pharmacokinetic drug interaction by comparing the steady-state pharmacokinetic characteristics of each arms after repeated administrating Lipilfen cap. 160mg and Livalo tab. 2mg through 3 period by separately or combinedly.

DETAILED DESCRIPTION:
To develop combination product of micronized fenofibrate plus pitavastatin, we would like to evaluate pharmacokinetic drug interaction by comparing the steady-state pharmacokinetic characteristics of each arms after repeated administrating Lipilfen cap. 160mg(micronized fenofibrate 160mg)by Dae Woong Pharma. and Livaro tab. 2mg (pitavastatin Ca 2mg) by Joong Wae Pharm. through 3 period by separately or combinedly.

ELIGIBILITY:
Inclusion Criteria:

1. Years 20-55
2. Body weight≥50kg and 18≤BMI≤29kg/m2
3. Volunteer

Exclusion Criteria:

1. Subject with serious active cardiovascular, respiratory, hepatology, renal, hematologic, gastrointestinal, immunologic, dermal, neurologic, or psychological disease or history of such disease
2. Subject with symptoms of acute disease within 28days prior to study medication dosing
3. Subject with known for history which affect on the absorption, distribution, metabolism or excretion of drug
4. Subject with clinically significant active chronic disease
5. Subject with any of the following conditions in laboratory test i. AST(aspartate aminotransferase) or ALT(alanine transferase) > upper normal limit × 1.5 ii. Total bilirubin > upper normal limit × 1.5 iii. renal failure with Creatinine clearance < 50mL/min iv. creatine phosphokinase > upper normal limit × 2
6. Positive test results for hepatitis B virus surface antigen, anti-hepatitis C virus antibody, venereal disease research laboratory test
7. Use of any prescription medication within 14 days prior to study medication dosing
8. Use of any medication such as over-the-counter medication including oriental medication within 7 days prior to study medication dosing
9. Subject with clinically significant allergic disease (except for mild allergic rhinitis and mild allergic dermatitis that are not needed to administer drug)
10. Subject with known for hypersensitivity reaction to fenofibrate, fenofibric acid or statin
11. gallbladder disease
12. Subject who experiences photo-allergy or photo-toxicity during administrating fibrates or ketoprofen
13. Subject with genetic deficiency such as galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption
14. Subject who is not albe to taking the institutional standard meal
15. Subject with whole blood donation within 60days, component blood donation within 20days
16. Subjects receiving blood transfusion within 30days prior to study medication dosing
17. Participation in any clinical investigation within 60days prior to study medication dosing
18. Continued excessive use of caffeine (caffeine > five cups/day), alcohol(alcohol>30g/day) and severe heavy smoker(cigarette > 10 cigarettes per day)
19. Subjects with decision of nonparticipation through investigator's review due to laboratory test results or other excuse such as non-responding to request or instruction by investigator

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Drug-Drug interaction evaluation (Cmax,ss, Cmin,ss, Tmax,ss) | just before dosing on 1st day and 4th day of each period and 0, 0.25, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48hr on final 5th dosing

SECONDARY OUTCOMES:
Number of participants with adverse events | Participants will be followed for the duration of study medication dosing days and hospital stay, and expected average of 3days and follow-up period for maximum 7 days from the discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea